CLINICAL TRIAL: NCT04931667
Title: A 3-Year, Multicenter, Open-Label Study Evaluating the Safety, Tolerability, and Efficacy of Intra-articular Lorecivivint in Subjects With Osteoarthritis of the Knee in a Real-World Setting (STRIDES-EXTRA)
Brief Title: 3-year, Open-Label Study Evaluating Safety, Tolerability, and Efficacy of Lorecivivint in Subjects With Osteoarthritis of the Knee
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to business reasons by Sponsor.
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SM04690-OA-17
Record Dates: First submitted 2021-06-04; First posted 2021-06-18 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Osteoarthritis of the Knee
Keywords: SM04690; Wnt pathway inhibitor; osteoarthritis; Biosplice Therapeutics, Inc.; Lorecivivint
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — lorecivivint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 0.07 mg Lorecivivint (Experimental): One intra-articular injection of 0.07 mg Lorecivivint in 2 ml vehicle in one or both knees as clinically indicated. Bilateral injection of 0.07 mg LOR are allowed.
  Interventions: Drug: Lorecivivint

INTERVENTIONS:
Drug: Lorecivivint — Healthcare professional-administered intra-articular (IA) injection into one or both knees as clinically indicated. Bilateral injections of 0.07 mg of LOR are allowed. IA injection performed on Day 1. Additional IA injections of LOR to same knee (with at least a 6 month separation) between Day 1 and Month 33.
  Other Names: SM04690

SUMMARY:
This study is designed as a 3-year, multicenter, open-label study evaluating the safety, tolerability, and efficacy of intra-articular (IA) Lorecivivint (LOR) in subjects with osteoarthritis of the knee in a real-world setting.

DETAILED DESCRIPTION:
At Day 1, after a screening period of up to 14 days, subjects will receive an IA injection of 0.07 mg LOR into one or both knees, followed by a 36-month evaluation period. Clinic visits will be scheduled at Day 1, and Months 3, 12, 24, and 36 [End of study (EOS)] or Early Termination (ET) for completion of all Patient Reported Outcome (PRO) measurements Western Ontario and McMaster University Arthritis Index (WOMAC), Knee Injury and Ostheoarthritis Outcome Score (KOOS), pain Numeric Rating Scale (NRS), Study Form (SF)-12, Patient Acceptable Symptom State Questionnaire (PASS), Work Productivity and Activity Impairment Questionnaire (WPAI)], functional tests [40-meter walk test and Time Up and Go (TUG) test at a subset of sites], and safety evaluations. On Day 1, the Charlson Comorbidity Index and Widespread Pain Index and Symptom Severity [WPI&SS] assessments will also be completed. A phone visit for safety follow-up will occur 4 weeks after the injection on Day 1. Subjects may also have Unscheduled Injection Visits for additional injections of LOR, glucocorticoid, or hyaluronic acid (HA). Following each injection, subjects will return to the clinic for 3-Month Post-Injection Follow-Up Visits, unless another visit has occurred between the injection and the 3-month post injection date. At these injection visits and 3-Month Post-Injection Follow-Up Visits, subjects will complete PRO measurements and functional tests (at a subset of sites).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 40 and 80 years of age, inclusive, in general good health apart from their knee OA
2. Femorotibial OA by standard American College of Rheumatology (ACR) criteria; knee OA is not to be secondary to any rheumatologic conditions (e.g., rheumatoid arthritis).
3. Pain compatible with knee OA for at least 26 weeks prior to the Screening Visit
4. Negative drug test for amphetamine, buprenorphine, cocaine, methadone, opiates, phencyclidine (PCP), propoxyphene, barbiturates, and benzodiazepine, unless any of these drugs are prescribed by a physician to treat a specific condition
5. Full understanding of the requirements of the study and willingness to comply with all study visits and assessments
6. Subjects must have read and understood the informed consent form (ICF), and must have signed and dated it prior to any study-related procedure being performed

Exclusion Criteria:

1. Pregnant women, breastfeeding women, and women who are not post-menopausal (defined as 12 months with no menses without an alternative medical cause) or permanently surgically sterile (includes hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) who have a positive or indeterminate pregnancy test result at Screening and Day 1
2. Women who are not post-menopausal or permanently surgically sterile who are sexually active, and who are not willing to use birth control during the study period
3. Any surgery (e.g., arthroscopy) in either knee within 26 weeks prior to Day 1
4. Intra-articular (IA) injection into either knee with a therapeutic aim including, but not limited to, hyaluronic acid, platelet-rich plasma (PRP), and stem cell therapies within 26 weeks prior to Day 1 or IA glucocorticoids within 12 weeks prior to Day 1
5. Any condition that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
6. Any comorbid condition that could affect study endpoint assessments of the knee, including, but not limited to, rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, gout or pseudogout, and fibromyalgia
7. Any contraindications for an IA injection in the knee(s) to be injected at Day 1 in the opinion of the Investigator

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | From Study Day 1 through Subject's last visit, Early Termination (ET) or End of Study (EOS), up to 36 months.
  AEs that occur during the study will be recorded. All AEs will be evaluated for severity, seriousness and causal relationship to study medication.

SECONDARY OUTCOMES:
Change from baseline in pain numeric rating scale (NRS) score for the knee | 3 months after each injection (planned and unscheduled) monitored throughout the study for up to 36 months
  Change from baseline in pain numeric rating scale (NRS) score for the knee. The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain.
Change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) physical function subscore (WOMAC Function) | 3 months after each injection (planned and unscheduled) monitored throughout the study for up to 36 months
  Change from baseline OA function in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) physical function subscore (WOMAC Function). The WOMAC is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with OA of the knee and hip, including pain, stiffness, and physical functioning of a target joint. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 4 (highest pain/highest stiffness/lowest function). The WOMAC Function subscore ranges from 0 to 68 (raw) and will be scaled 0 to 100 for reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, MD, Study Director — Biosplice Therapeutics, Inc.
Locations (4):
- United States (4):
  - Research Site, Tucson, Arizona
  - Research Site, Winter Park, Florida
  - Research Site, Oak Brook, Illinois
  - Research Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No